CLINICAL TRIAL: NCT06422663
Title: A Prospective, Observational, Multicentre Study To Evaluate The Treatment Pattern Of Moderate-to-Severe Asthma Patients In China
Brief Title: A Study To Evaluate The Treatment Pattern Of Moderate-to-Severe Asthma Patients In China
Acronym: PRESENT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00198
Record Dates: First submitted 2024-03-19; First posted 2024-05-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Moderate-to-Severe Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate-to-Severe Asthma: enroll 500 subjects

SUMMARY:
This is a Prospective, Observational, Multicentre Study to describe treatment pattern changes of uncontrolled moderate-to-severe asthma patients in China. Sponsor by Astrazeneca Investment(China) Co., LTD.

DETAILED DESCRIPTION:
This is a prospective, observational, multicentre study. Approximately 500 moderate-to-severe asthma patients from 30 sites across China. Patients will be treated following routine clinical practice. Study measures will be collected at week 0, week 12 and week 24.

The primary objective of PRESENT study is to describe treatment pattern changes of uncontrolled moderate-to-severe asthma patients in China.

ELIGIBILITY:
Inclusion Criteria:

1. Physician-confirmed asthma diagnosis with documented evidence of variable expiratory airflow limitation (e.g., from bronchodilator reversibility testing or other tests)
2. Written informed consent
3. Moderate-to-severe asthma (asthma patients with treatment of GINA Step 3-5)
4. Age 12 years old and above

Exclusion Criteria:

1. Previous diagnosis of chronic obstructive pulmonary disease (COPD) or other clinically relevant chronic respiratory disease other than asthma
2. Received an investigational therapy for asthma, allergy, atopic disease, or eosinophilic disease as part of a clinical trial during the 6 months prior to enrolment. (Once enrolled in the PRESENT Study, patients should not enrol in any investigational trials.)
3. Any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate in the study
4. Disease or condition other than asthma that requires treatment with systemic or oral steroids
5. Patients with poor inhaler skills and adherence

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moderate-to-Severe Asthma Patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Proportion of uncontrolled patients with treatment modification, which is indicated by maintenance drug dosage change, switch, add-on, discontinue from week 0 to week 24 | week 0, week 12 and week 24.
  To describe treatment modification of uncontrolled moderate-to-severe asthma patients in China.

SECONDARY OUTCOMES:
Ashma disease burden: Exacerbation rate | week 0, week 12 and week 24
  To describe disease burden of moderate-to-severe-asthma patients and to describe by different subgroups. To describe disease burden and treatment patterns by stratification of baseline EOS and baseline eosinophilic phenotype at week 0,12&24. To describe disease burden and treatment patterns by baseline asthma severity(moderate or severe) at each follow-up assessment. To describe disease burden and treatment patterns by regions (south, west, east, north, central)
Proportions of severe asthma (GINA 2023 & CN 2020 guideline) at baseline & each follow-up assessment | week 0, week 12 and week 24
  To describe the proportion of severe asthma among all patients according to GINA 2023 & CN 2020 guidelines
Levels of bEOS at each follow-up assessment. Proportions of eosinophilic phenotype | week 0, week 12 and week 24
  To describe EOS levels and proportion of eosinophilic phenotype patients at week 0,12&24
Asthma-related emergency visit. | week 0, week 12 and week 24
  To describe healthcare utilization by baseline asthma severity (moderate or severe)
Ashma disease burden: Asthma Control Test | week 0, week 12 and week 24
  To describe disease burden of moderate-to-severe-asthma patients and to describe by different subgroups. To describe disease burden and treatment patterns by stratification of baseline EOS and baseline eosinophilic phenotype at week 0,12&24. To describe disease burden and treatment patterns by baseline asthma severity(moderate or severe) at each follow-up assessment. To describe disease burden and treatment patterns by regions (south, west, east, north, central)
Ashma disease burden: Lung function (FEV1) | week 0, week 12 and week 24
  To describe disease burden of moderate-to-severe-asthma patients and to describe by different subgroups. To describe disease burden and treatment patterns by stratification of baseline EOS and baseline eosinophilic phenotype at week 0,12&24. To describe disease burden and treatment patterns by baseline asthma severity(moderate or severe) at each follow-up assessment. To describe disease burden and treatment patterns by regions (south, west, east, north, central)
Asthma disease burden: Treatment patterns | week 0, week 12 and week 24
  To describe disease burden and treatment patterns by stratification of baseline EOS and baseline eosinophilic phenotype at week 0,12&24. To describe disease burden and treatment patterns by baseline asthma severity(moderate or severe) at each follow-up assessment. To describe disease burden and treatment patterns by regions (south, west, east, north, central)
Asthma-related outpatient visit. | week 0, week 12 and week 24
  To describe healthcare utilization by baseline asthma severity (moderate or severe)
Asthma-related hospitalization: Length of stay, Invasive and non-invasive ventilator use. | week 0, week 12 and week 24
  To describe healthcare utilization by baseline asthma severity (moderate or severe)
Asthma-related diagnostic tests (X-ray, CT scan, et al.) | week 0, week 12 and week 24
  To describe healthcare utilization by baseline asthma severity (moderate or severe)

OTHER OUTCOMES:
Frequency of adverse events | week 0, week 12 and week 24
  To summarize the safety data, including frequency of adverse events
Percentage of adverse events. | week 0, week 12 and week 24
  To summarize the safety data, including percentage of adverse events.
Frequency of serious adverse events. | week 0, week 12 and week 24.
  To summarize the safety data, including frequency of serious adverse events.
Percentage of serious adverse events. | week 0, week 12 and week 24
  To summarize the safety data, including percentage of serious adverse events.

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dingzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Liuchow
  - Research Site, Lu'an
  - Research Site, Luzhou
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Qingdao
  - Research Site, Quanzhou
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Tiaobingshan
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yongzhou
  - Research Site, Zhangjiagang
  - Research Site, Zhengzhou
  - Research Site, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  URL: https://vivli.org/
URL: https://vivli.org/